CLINICAL TRIAL: NCT02635646
Title: Efficacy of a Family and Interdisciplinary Intervention to Prevent Diabetes, and Effect on Family Profiles of Insulin Secretion and Insulin Resistance in Patients With Prediabetes
Brief Title: Interdisciplinary and Family Intervention to Prevent Type 2 Diabetes
Acronym: CARE-in-DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: University of Texas (Other); National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Rodolfo Guardado Mendoza, Titular Profesor A, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UG 1/2014
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family and interdisciplinary approach (Experimental): Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Interventions: Other: Family and interdisciplinary approach
- individual approach (Active Comparator): individual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  Interventions: Other: individual approach

INTERVENTIONS:
Other: Family and interdisciplinary approach — Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  Arms: Family and interdisciplinary approach
Other: individual approach — individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  Arms: individual approach

SUMMARY:
The purpose of the study is to evaluate the effect of a family and interdisciplinary approach on individual and family insulin resistance and insulin secretion in patients with prediabetes.

DETAILED DESCRIPTION:
This a randomized clinical trial designed to evaluate the efficacy of the following treatments:

1. Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
2. Individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months

To improve individual and family insulin resistance and insulin secretion in patients with prediabetes.

Patients will have a follow-up visit every month in the Metabolic Research Laboratory at the University of Guanajuato, Mexico, and will have a fasting measurement of lipids, glucose and insulin every 3 months, as well as 2h oral glucose tolerance test (OGTT) at basal, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prediabetes (Fasting glucose 100-125mg/dl and/or 2h post OGTT glucose 140-199mg/dl)
* Family of patients with prediabetes (in case of the patients that are randomized to FAMILY APPROACH)
* Signing of the inform consent

Exclusion Criteria:

* Type 2 diabetes
* Pregnancy
* Liver disease
* Renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Guardado, Dr, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  56 patients were included in this group
- Individual Approach: Iindividual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  Individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  58 patients were included in this group
Period: Overall Study
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Started | 57 | 65
Completed | 32 | 39
Not Completed | 25 | 26
Not completed — Lost to Follow-up | 24 | 25
Not completed — Pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
- Individual Approach: Iindividual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  Individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
- Total: Total of all reporting groups
Arm/Group | Family and Interdisciplinary Approach | Individual Approach | Total
Number analyzed (Participants) | 57 | 65 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13) | 46 (12) | 44 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 25 | 34 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 65 | 122
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Individual Insulin Resistance and Insulin Secretion
Description: Whole body insulin sensitivity as determined by the Matsuda Index was calculated using the following formula: 10,000 divided by the square root of (FPI* FPG) * (xGPC* xIPC) Where FPI is fasting plasma insulin expressed as uU/ml, FPG is fasting plasma glucose expressed as mg/dL, xGPC is mean plasma glucose concentration after the load and xIPC is the mean insulin concentration after the load. Values calculated on samples taken at 0, 30, 60, 90 and 120 minutes of a 2 hour OGTT. Values typically range from 0 to 12 units with higher scores indicating better insulin sensitivity (better result). A value of 2.5 or less is indicative of low insulin sensitivity (worst result).
Time Frame: 6 months
Population: The analysis was performed only in patients completing the 6 month follow-up, since there were patients lost during the follow-up by drop-outs
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  57 patients were included in this group
- Individual Approach: individual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  65 patients were included in this group
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Number analyzed (Participants) | 42 | 48
score on a scale | 4.9 (3.5) | 4.8 (2.6)
Statistical Analysis 1: Comparison: Family and Interdisciplinary Approach vs Individual Approach; Test type: Other — T test for mean comparisons between independent groups; p = 0.844, t-test, 2 sided — Significant p value less than 0.05

2. Primary Outcome: Individual Insulin Resistance and Insulin Secretion
Description: Whole body insulin sensitivity as determined by the Matsuda Index was calculated using the following formula: 10,000 divided by the square root of (FPI* FPG) * (xGPC* xIPC) Where FPI is fasting plasma insulin expressed as uU/ml, FPG is fasting plasma glucose expressed as mg/dL, xGPC is mean plasma glucose concentration after the load and xIPC is the mean insulin concentration after the load. Values calculated on samples taken at 0, 30, 60, 90 and 120 minutes of a 2 hour OGTT. Values typically range from 0 to 12 units with higher values indicating better insulin sensitivity (better result, the higher the value the better the result of this variable). A value of 2.5 or less is indicative of low insulin sensitivity (worst result).
Time Frame: 12 months
Population: Only the patients that completed the 12-months follow-up were included in this analysis, since some patients drop-out from the study before the 12-months follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  57 patients started in this group, but only 32 completed the 12-month follow-up
- Individual Approach: individual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  65 patients started in this group, but only 39 completed the 12-month follow-up
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Number analyzed (Participants) | 32 | 39
score on a scale | 4.7 (3.5) | 4.9 (3.0)
Statistical Analysis 1: Comparison: Family and Interdisciplinary Approach vs Individual Approach; Test type: Other; p = 0.624, t-test, 2 sided

3. Secondary Outcome: Family Insulin Resistance and Insulin Secretion (Matsuda Index Measured in the Relatives of the Patients)
Description: Whole body insulin sensitivity as determined by the Matsuda Index as calculated using the following formula: 10,000 divided by the square root of (FPI* FPG) * (xGPC* xIPC) Where FPI is fasting plasma insulin expressed as uU/ml, FPG is fasting plasma glucose expressed as mg/dL, xGPC is mean plasma glucose concentration after the load and xIPC is the mean insulin concentration after the load. Values calculated on samples taken at 0, 30, 60, 90 and 120 minutes of a 2 hour OGTT. Values typically range from 0 to 12 units with higher scores indicating better insulin sensitivity (the higher the value the better the result). A value of 2.5 or less is indicative of low insulin sensitivity (worst result).
Time Frame: 12 months
Population: Matsuda Index measured in the relatives of the patients at the end of the study (12 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  68 patients were included in this group, but only 23 completed the 12-month follow-up
- Individual Approach: Iindividual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  Individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  33 patients were included in this group, but only 7 completed the 12-month follow-up
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Number analyzed (Participants) | 23 | 7
score on a scale | 5.5 (2.6) | 4.6 (3.5)
Statistical Analysis 1: Comparison: Family and Interdisciplinary Approach vs Individual Approach; Test type: Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Weight
Description: Weight in the relatives of the patients
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Number analyzed (Participants) | 23 | 7
kg | 65.4 (16.8) | 75.0 (16.0)
Statistical Analysis 1: Comparison: Family and Interdisciplinary Approach vs Individual Approach; Test type: Other; p = 0.516, t-test, 2 sided

5. Secondary Outcome: 2h OGTT Glucose
Description: Measurement of 2h post OGTT glucose
Time Frame: 6 and 12 months
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Family and Interdisciplinary Approach: Family and interdisciplinary approach: Patients in this group will receive a Family and interdisciplinary approach that includes nutritional, physical activity and psychological counseling + metformin 850mg twice at day for 12 months
  Family and interdisciplinary approach: Family and interdisciplinary approach that includes:
  1. nutritional counseling,
  2. physical activity counseling,
  3. psychological counseling,
  4. metformin 850mg twice at day for 12 months All this with the purpose to improve insulin resistance and insulin secretion in patients with prediabetes. Patients must attend a monthly session together with his family where they will receive the nutritional, physical activity and psychological counseling.
  57 patients were included in this group, but only 32 patients completed the 12-month follow-up
- Individual Approach: individual approach: Patients in this group will receive individual approach that includes nutritional and physical activity counseling + metformin 850mg twice at day for 12 months
  individual approach: Individual approach that includes:
  1. nutritional and physical activity counseling in individual appointments,
  2. metformin 850mg twice at day for 12 months, All this with the purpose to improve insulin resistance and insulin secretion. The patients must attend a monthly follow-up individually.
  65 patients were included in this group, but only 39 patients completed the 12-month follow-up
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Number analyzed (Participants) | 32 | 39
mg/dl
  2h Glucose at 6 months | 135 (35) | 131 (45)
  2h Glucose at 12 months | 142 (33) | 127 (33)
Statistical Analysis 1: Comparison: Family and Interdisciplinary Approach vs Individual Approach; Test type: Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during 1 year
Description: Non serious adverse evens were expected to occur during this study
Arm/Group | Family and Interdisciplinary Approach | Individual Approach
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/65
Other Adverse Events (participants affected / at risk) | 0/57 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No